CLINICAL TRIAL: NCT04761991
Title: Comparison of Cardiovascular Magnetic Resonance and Computed Tomography With Fractional Flow Reserve in the Diagnosis of Suspected Coronary Artery Disease
Brief Title: CMR Versus CT in Coronary Artery Disease
Acronym: CONCORD
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: HeartFlow, Inc. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Oxford (Other); University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: 0726/258996; 1ZIAHL006242-02 (NIH)
Record Dates: First submitted 2020-12-17; First posted 2021-02-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease
Keywords: MRI; CT-FFR; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: CMR and CTCA with CT-FFR — multi-parametric CMR assessment and CT coronary angiography with FFR assessment

SUMMARY:
CONCORD is a prospective observational study evaluating the diagnostic accuracy of cardiovascular magnetic resonance (CMR) and computed tomography with fractional flow reserve (CT-FFR) in patients with suspected coronary artery disease, using invasive fractional flow reserve (FFR) as the reference standard.

DETAILED DESCRIPTION:
In patients with suspected coronary artery disease (CAD), CT coronary angiography (CTCA) provides excellent sensitivity and negative predictive value, enabling the safe exclusion of significant CAD. However, its positive predictive value remains suboptimal (c.50%). Undertaking additional CT-FFR improves specificity and positive predictive value, reducing unnecessary invasive coronary angiography. It has been established that CMR perfusion imaging offers excellent diagnostic accuracy for the identification of functionally significant coronary artery disease. The diagnostic performance of qualitative CMR perfusion assessment may be further enhanced by additional quantitative assessment. The purpose of this prospective observational study is to evaluate the diagnostic performance of all three modalities (CT-FFR and qualitative and quantitative CMR perfusion imaging), involving 300 patients with suspected coronary artery disease referred for invasive coronary angiography. A subset of 167 subjects will undergo an additional accelerated CMR scan for comparison. Invasively measured fractional flow reserve (FFR) will serve as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Referred for invasive coronary angiography for investigation of chest pain

Exclusion Criteria:

* Recent acute coronary syndrome (< 6 months)
* Previous coronary artery bypass grafting
* Severe claustrophobia
* Absolute contraindications to CMR - those with MR conditional or safe devices will be included
* Second-/third-degree atrioventricular block
* Severe chronic obstructive pulmonary disease
* Moderate-severe asthma
* Estimated glomerular filtration rate <30 ml/min/1.73m2
* Women who are pregnant, breast-feeding or of child-bearing potential( premenopausal women)
* Contraindication to iodinated contrast
* Participation in a research study involving an investigational product in the past 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected coronary artery disease referred for invasive coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
1. Diagnostic performance of CMR and CT-FFR | 6 weeks
  Diagnostic accuracy of CMR perfusion imaging (quantitative and qualitative analysis) and CT-FFR to determine the presence/absence of significant coronary artery disease at the subject level when compared with invasive FFR.

SECONDARY OUTCOMES:
1. Diagnostic performance of CMR and CT-FFR | 6 weeks
  1. Sensitivity and specificity of CMR perfusion imaging (quantitative and qualitative analysis) and CT-FFR to determine the presence/absence of significant coronary artery disease at the subject level when compared with invasive FFR.
2. Diagnostic performance of CMR and CT-FFR | 6 weeks
  2. Diagnostic accuracy, sensitivity and specificity of CMR perfusion imaging (quantitative and qualitative analysis) and CT-FFR to determine the presence/absence of significant coronary artery disease at the vessel level when compared with invasive FFR.
3. Diagnostic performance of CMR T1 mapping | 6 weeks
  Diagnostic accuracy, sensitivity and specificity of CMR T1 mapping using invasive FFR as the reference standard (per patient and per vessel levels).
4. Diagnostic performance of hybrid imaging | 6 weeks
  Diagnostic accuracy, sensitivity and specificity of hybrid CMR/CT-FFR using invasive FFR as the reference standard (per patient and per vessel levels).
Diagnostic performance of strain assessment | 6 weeks
  5. Diagnostic accuracy, sensitivity and specificity of CMR strain assessment (global/segmental longitudinal/circumferential strain, mechanical dispersion) using invasive FFR as the reference standard (per patient and per vessel levels).
6. Cost analysis | 2 years
  Cost analysis to assess the long term costs of the different diagnostic testing strategies. Healthcare costs for each testing strategy - data on resource use (staff time, scan duration, hospital days and clinic visits) will be collected during the study period.
7. Clinical endpoints | 2 years
  Prediction by imaging modalities of clinical endpoints (subsequent percutaneous and/or surgical revascularisation, admissions with acute coronary syndrome and cerebrovascular accident, all-cause mortality).
8. Subjective experience | 1 day
  Subjective patient scan experience for CMR and CTCA.
9. Time duration of each scan/scan component. | 1 day
  Duration of each scan/scan component.
10. Image quality | 1 day
  Image quality of each scan/scan component, assessed visually on a 4-point score - excellent (3), good (2), moderate (1) and poor (0).

CONTACTS AND LOCATIONS:
Locations (1):
- Glenfield Hospital, Leicester, Leics, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shergill S, Elshibly M, Parke KS, England R, Wormleighton JV, Das I, Gulsin GS, Hothi SS, Heggie R, Wu O, Kellman P, McIntosh A, McConnachie A, Ladwiniec A, McCann GP, Arnold JR. Cardiovascular magnetic resonance versus coronary computed tomography angiography with fractional flow reserve for diagnosing obstructive coronary artery disease in higher risk patients: rationale and design of CONCORD-A prospective, single-center diagnostic accuracy study. J Cardiovasc Magn Reson. 2025 Aug 14;28(1):101939. doi: 10.1016/j.jocmr.2025.101939. Online ahead of print. PMID 40818667